CLINICAL TRIAL: NCT05402917
Title: Comparison of Post-operative Analgesia Efficacy of Erector Spina Plan Block (ESPB) and Thoracic Epidural Analgesia (TEA) in Patients Undergoing Lobectomy With Thoracotomy Incision
Brief Title: Comparison of the Efficacy of Erector Spina Plane Block and Thoracic Epidural Analgesia After Thoracotomy
Acronym: ESPBTEAPAIN
Status: Completed | Type: Observational
Sponsor: Mesut Aslan (Other)
Responsible Party: Sponsor-Investigator, Mesut Aslan, Asistant Doctor, Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital
Organization: Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other)
Other Study IDs: espVStea
Record Dates: First submitted 2022-05-25; First posted 2022-06-02 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Pain, Postoperative
Keywords: ESPB; TEA; THORACOTOMY
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thoracic Epidural Analgesia (TEA): For patients undergoing TEA is done under general anesthesia after surgery procedure.Once the catheter is secured, a bolus dose of 15 ml of 0.25% bupivacaine will be administered as an epidural injection through the catheter, followed by a continuous infusion of 0.125% bupivacaine at a rate of 0.1 mL/kg/h for the postoperative 24-hour period.
- Erector Spina Plan Block (ESPB): For patients undergoing ESPB is done under general anesthesia after surgery procedure.A bolus dose of 15 mL of 0.25% bupivacaine will be administered from the inserted catheter. Subsequently, 0.125% bupivacaine will be given continuously at a rate of 0.1 mL/kg/h for up to 24 hours post-operatively.
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Interfascial plane (area) blocks are blocks in which the local anesthetic agent is injected into the potential area between the two fasciae. The ESPB we used in our study is a member of interfascial plane blocks. The erector is applied between the spinal muscle and the transverse process, spreading the drug from the injection site to both cranial and caudal. Unlike other defined interfascial plane blocks, ESPB can show paraspinal block characteristics since the injection site is above the transverse process.
  Groups: Erector Spina Plan Block (ESPB)

SUMMARY:
In patients who undergoing lobectomy with thoracotomy incision, the effectiveness of erector spina plane block in post-operative analgesia management is at least as much as thoracic epidural anesthesia.

DETAILED DESCRIPTION:
Observational recording of the data was planned by dividing the patients who met the internal criteria of the study and whose written and verbal consents were obtained for the study, into two groups as the patients applied ESPB or TEA. ESPB and TEA are applied to patients in our clinic depending on the preference of the physician. The routine procedures in ESPB and TEA are described in groups part. For this study, no procedure or intervention other than this routine will be performed, and the research will be conducted observationally.

Anesthesia induction for both groups will be performed with standard monitors, electrocardiogram, peripheral oxygen saturation probe and non-invasive automatic blood pressure/invasive arterial monitoring in the operating room. Anesthesia induction will be performed with 2 mg/kg propofol, 2 mcg/kg fentanyl and 0.6 mg/kg rocuronium with 1.5 mg/kg IV lidocaine, followed by double lumen endotracheal intubation and positive pressure mechanical ventilation with controlled positive 50% inspired oxygen. Ventilation parameters will be adjusted to keep end-tidal carbon dioxide around 35 mmHg. Anesthesia will be maintained with end-tidal sevoflurane 0.7-1.5 minimum alveolar concentration (adjusted for hemodynamics) 0.15 mg/kg rocuronium and 0.05-0.2 mcg/kg/min remifentanil (adjusted for hemodynamics). Acetaminophen (1 g paracetamol) IV will be administered to all patients 30 minutes before the end of surgery.

Blood pressure, peripheral oxygen saturation, heart rate, end-pulmonary carbon dioxide value and mac value of the patients will be recorded before and after block application, before and after anesthesia induction, every 15 minutes in the first hour and every 30 minutes after the first hour. Patients will be extubated with 0.03 mg/kg atropine and 0.07 mg/kg neostigmine at the end of surgery. Hemodynamic and resting Visual Analogue Scale (VAS) values for both groups taken to the post-operative intensive care unit will be recorded by nurse or anesthesia assistant at 0,2, 4, 8, 16 and 24 hours after their admittance to the intensive care unit. In combination with the numerical pain scale, the Wong-Baker face pain scale (FS) will be used for the postoperative pain assessment of the patient. The pain assessment form will have six faces representing pain along with numbers 0 to 10, with 0 for no pain and 10 for being unbearable pain. Post-operative nausea, vomiting and any complications related to the block will be reported. Patients in the two groups will be evaluated with the VAS score for the pain they describe and record; VAS 0-4 will be classified as mild, VAS 5-7 as moderate, VAS 8-10 as severe pain. In patients with VAS >4, additional analgesia will be given with IV non-steroidal anti-inflammatory drugs (20 mg tenoxicam); after 30 minutes, VAS scoring will be evaluated again and IV tramadol 2 mg/kg (not to exceed a maximum of 100 mg once and not to exceed a maximum of 400 mg daily) will be administered in addition to patients with VAS>4. Additional analgesia amounts and hours used will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Lobectomy planned with thoracotomy incision;
* Adult aged 18-75;
* American Society of Anesthesiology(ASA) score1-3.

Exclusion Criteria:

* Obesity (BMI greater than 35 kg/m2)
* Local infection at the injection site,
* Presence of known coagulopathy
* Bone or brain metastasis
* Having impaired liver or kidney function
* Patients who cannot evaluate VAS as cognitive function
* Patients who cannot use the Patient-Controlled Analgesia (PCA) pump as a -cognitive function
* History of chronic pain medication use
* Allergy to the drugs to be used in the study
* Withdrawing consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing lobectomy with thoracotomy incision
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) Change | The first 24 hours postoperatively is the end time for primary outcome measurement.Visual Analogue Scale (VAS) change values for both groups will be recorded at 0, 2, 4, 8, 16 and 24 hours after their admittance to the intensive care unit.
  The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Wong-Baker Face Pain Scale (FS) Change | The first 24 hours postoperatively is the end time for primary outcome measurement.Wong-Baker Face Pain Scale(FS) values change for both groups will be recorded at 0, 2, 4, 8, 16 and 24 hours after their admittance to the intensive care unit.
  The scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable.

SECONDARY OUTCOMES:
Hemodynamic Values Change | The first 24 hours postoperatively is the end time for secondary outcome measurement. Hemodynamic values change for both groups will be recorded at 0, 2, 4, 8, 16 and 24 hours after their admittance to the intensive care unit.
  Blood Pressure: mmhg Heart Rate: beat/minute
Pulse Oximetry(SpO2) Change | The first 24 hours postoperatively is the end time for secondary outcome measurement. Pulse Oximetry(SpO2) change values for both groups will be recorded at 0, 2, 4, 8, 16 and 24 hours after their admittance to the intensive care unit.
  %0-100.
Postoperative Nausea and Vomiting(PONV) Change | The first 24 hours postoperatively is the end time for secondary outcome measurement. Postoperative nausea or vomiting change for both groups will be recorded at 0, 2, 4, 8, 16 and 24 hours after their admittance to the intensive care unit.
  If nausea and vomiting exist, it will be recorded as '1', if not, it will be recorded as '0'.
Nonsteroidal Anti-inflammatory Drug Usage Need Change | The first 24 hours postoperatively is the end time for secondary outcome measurement. Nonsteroidal anti-inflammatory drug usage need change for both groups will be recorded at 0, 2, 4, 8, 16 and 24 hours after their admittance to the intensive care unit.
  If nonsteroidal anti-inflammatory drug is used: 1 If nonsteroidal anti-inflammatory drug is not used: 0
Opioid Drug Usage Need Change | The first 24 hours postoperatively is the end time for secondary outcome measurement. Opioid drug usage need change for both groups will be recorded at 0, 2, 4, 8, 16 and 24 hours after their admittance to the intensive care unit.
  If opioid drug is used: 1 If opioid drug is not used: 0

CONTACTS AND LOCATIONS:
Locations (1):
- Dr.Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)